CLINICAL TRIAL: NCT05789966
Title: The Effect of Communicating Genetic Risk of Coronary Heart Disease and Wearable Technologies On Wearable-Device-Measured Behavioral Outcomes in East Asians: Protocol of a Randomized Controlled Trial
Brief Title: Fullscale_Intervention Study: Genetic Risk Communication in Coronary Heart Disease and Wearables
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kim, Youngwon, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Fullscale_CHD_RCT
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Fitness Trackers; Sedentary Time; Genetic Predisposition to Disease; Coronary Heart Disease
Keywords: Coronary Heart Disease; Genetic risk; Sedentary Time; Wearable Technology; Randomized Controlled Trial
MeSH Terms: conditions — Sedentary Behavior; Genetic Predisposition to Disease; Coronary Disease

STUDY DESIGN:
Intervention Model Description: parallel-group, open randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Staff without knowledge of participant information will create a computer-generated list that consists of blocks of six that contain two of each of the three groups per block in a random order. The randomisation list will be incorporated into a computer program that our staff will use for enrolment and automated random assignment of participants. Group allocation will be concealed from study staff until the 7-day pre-intervention period begins (to allow preparation of genetic risk estimates and/or calculate Fitbit step goals from baseline data) and concealed from participants until the intervention begins. Given the nature of the interventions, it is impossible for participants to be blinded to their group allocation; however, research staff analysing participants' deidentified data will remain blinded to participant group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group will receive a Fitbit device
- Intervention Group - Genetic Risk Estimate+health coaching (Experimental): Genetic: Genetic Risk Estimate The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for CHD as well as a dichotomized genetic risk category: 'increased genetic risk' (if their genetic risk is higher than the average population risk) or 'no increased genetic risk' (if their genetic risk is not higher than the average population risk). Health coaching will be incorporated as well.
  Interventions: Genetic: Genetic Risk Estimate+Health Coaching; Device: Genetic Risk Estimate + Fitbit Functions+Health Coaching
- Intervention Group - Genetic Risk Estimate + Fitbit Functions+health coaching (Experimental): Device: Genetic Risk Estimate + Fitbit Functions The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for CHD as well as a dichotomized genetic risk category: 'increased genetic risk' or 'no increased genetic risk'.
  The two unique Fitbit functions are step goal setting and prompts. Individualized daily step goals will be set to be 10% higher than participants' own baseline Fitbit step counts. The 'Reminder To Move' function of Fitbit will be used as a prompt to remind participants to reduce sedentary time and walk at least 250 steps/hour within a specified timeframe (i.e., from 9am to 10pm in the proposed research). If the user has not accumulated at least 250 steps/hour, a reminder (for example, 150 steps to go) will appear on the Fitbit screen at 10 minutes before the hour (for example, at 10:50 a.m.) and cause the device to vibrate. Health coaching will be incorporated as well.
  Interventions: Device: Genetic Risk Estimate + Fitbit Functions+Health Coaching

INTERVENTIONS:
Genetic: Genetic Risk Estimate+Health Coaching — The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for CHD as well as a dichotomized genetic risk category: 'increased genetic risk' (if their genetic risk is higher than the average population risk) or 'no increased genetic risk' (if their genetic risk is not higher than the average population risk). Health coaching will be incorporated through phone or Zoom calls to provide an explanation of each participant's own genetic risk of CHD as well as lifestyle modification measures.
  Arms: Intervention Group - Genetic Risk Estimate+health coaching
Device: Genetic Risk Estimate + Fitbit Functions+Health Coaching — Intervention: Device: Genetic Risk Estimate + Fitbit Functions The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for CHD as well as a dichotomized genetic risk category: 'increased genetic risk' or 'no increased genetic risk'.
  The two unique Fitbit functions are step goal setting and prompts. Individualized daily step goals will be set to be 10% higher than participants' own baseline Fitbit step counts. The 'Reminder To Move' function of Fitbit will be used as a prompt to remind participants to reduce sedentary time and walk at least 250 steps/hour within a specified timeframe (i.e., from 9am to 10pm in the proposed research). If the user has not accumulated at least 250 steps/hour, a reminder (for example, 150 steps to go) will appear on the Fitbit screen at 10 minutes before the hour (for example, at 10:50 a.m.) and cause the device to vibrate. Health coaching will be incorporated as well
  Arms: Intervention Group - Genetic Risk Estimate + Fitbit Functions+health coaching; Intervention Group - Genetic Risk Estimate+health coaching

SUMMARY:
Background: This study aims to determine the effects of communicating genetic risk for Coronary Heart Disease (CHD) alone or in combination with goal setting and prompts from a wearable device on objectively measured sedentary time (ST) in East Asians. It is hypothesized that this combination will lead to significant favorable changes in objectively ST, and that such changes will be more likely to be sustained over 6-month follow-up.

Methods: In a parallel group, randomized controlled trial, a total 414 individuals of East Asians aged over 60years will be allocated into one of three groups: 1 control and 2 intervention groups. Blood samples will be used for estimation of CHD genetic and analysis of metabolic risk markers. Genetic risk for CHD will be estimated based on recently identified 79 SNPs (associated with CHD for East Asians) using an established methodology. Questionnaires and physical measurement will be administered at Before and after the 12-month intervention and at 6-month follow-up. Each group will receive a Fitbit device. Both intervention groups will be given CHD genetic risk estimates along with lifestyle advice but one of them will additionally use Fitbit's step-goal setting and prompt functions. The primary outcome is objectively measured sedentary time. Secondary outcomes include objectively measured MVPA, calories burned, and five intermediate metabolic risk markers (total cholesterol/HDL-C/LDL-C/triglycerides).

ELIGIBILITY:
Inclusion Criteria:

* East Asian ancestry
* Do not meet the WHO-recommended levels of PA (i.e., ≥150 minutes/week of moderate-intensity PA, ≥75 minutes/week of vigorous-intensity PA, or an equivalent combination of the two; determined through the IPAQ-Short Form).

Exclusion Criteria:

* Previously diagnosed with CHD, and/or participation in another exercise-intervention study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in ST (average, in minutes/day) between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, 12-month post-intervention, 6-month follow-up
  ST (average, in minutes/day) will be objectively measured by the Fitbit tracker.

SECONDARY OUTCOMES:
Changes in five activity indicators (steps, 'sedentary minutes', 'lightly active minutes', calories burn, and sleep time) | Baseline, 12-month post-intervention, 6-month follow-up
  steps, sedentary minutes, lightly active minutes, calories burn, and sleep time will be objectively measured by the Fitbit tracker.
Changes in four CHD markers (total cholesterol/HDL-C/LDL-C/triglycerides) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the four key markers for CHD
Changes in hand grip strength between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Hand grip strength (in kilograms) will be measured using the Jamar Hydraulic Hand Dynamometer, which has good reliability and reproducibility.
Changes in systolic/diastolic blood pressure between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Systolic/diastolic blood pressure will be measured using a digital automatic sphygmomanometer
Changes in Self-reported Physical Activity between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Fruit and Vegetable Consumption between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Smoking Status between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Psychological Status between baseline and Immediate post-intervention, between baseline and 12-month post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 12-month post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Youngwon Kim, Dr, Principal Investigator — The University of Hong Kong